CLINICAL TRIAL: NCT02210182
Title: A Phase I Clinical Study on the Hepatic Uptake, Pharmacokinetics, Safety and Tolerance of a New Oral Pentamidine Formulation in Hepatocellular Carcinoma Subjects Undergoing Thermal Ablation
Brief Title: A Phase I Clinical Study on a New Oral Pentamidine Formulation in Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncozyme Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCZ103-300-1401
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Oral Pentamidine; Endo-exonuclease
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Pentamidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral pentamidine (Experimental): Oral pentamidine given at 300 mg, 600 mg, 900 mg or 1200 mg QD x 3 consecutive days
  Interventions: Drug: Oral Pentamidine
- Placebo (Placebo Comparator): Placebo given at 300 mg, 600 mg, 900 mg or 1200 mg QD x 3 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Pentamidine — Oral pentamidine given at 300 mg, 600 mg, 900 mg or 1200 mg QD x 3 consecutive days
  Other Names: VLX103
  Arms: Oral pentamidine
Other: Placebo — Placebo given at 300 mg, 600 mg, 900 mg or 1200 mg QD x 3 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate on the Hepatic Uptake, Pharmacokinetics, Safety and Tolerance of a New Oral Pentamidine Formulation in Hepatocellular Carcinoma Subjects Undergoing Thermal Ablation

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, sequential-group administration of a new oral pentamidine formulation to investigate its hepatic uptake, pharmacokinetics, safety and tolerance in subjects with hepatocellular carcinoma who undergoes thermal ablation procedure

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects
2. 18 years of age or older
3. Radiologically established diagnosis of hepatocellular carcinoma (HCC) with tumor diameter ≤ 5 cm
4. Suitable for and scheduled to undergo thermal ablation as treatment
5. Have a Barcelona score of 0 or A
6. Have a Child Pugh score of A or B
7. Legally and mentally able to give informed consent to participate in the study
8. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects of the trial prior to enrolment
9. Willingness and ability to comply with scheduled visits and trial procedures

Exclusion Criteria:

1. Presence of uncontrolled diabetes, defined as glycated hemoglobin (Hb1Ac) ≥ 8.0
2. History of clinically significant hypoglycaemia, with fasting blood glucose < 3 mmol/L within 3 months prior to signature of ICF
3. Presence of clinically significant renal impairment, defined as a creatinine clearance < 60 mL/min
4. Systolic Blood Pressure < 100 mm Hg (if deemed clinically significant by the treating physician)
5. Current or recent (< 2 years) history of pancreatitis
6. International Normalised Ratio (INR) > 1.5 or presence of severe coagulation disorders (vg but limited to prothrombin activity < 40% or a platelet count of < 40,000 / mm3)
7. Presence of known vascular invasion, bile duct invasion or extrahepatic metastasis
8. Presence of portal venous thrombosis
9. Concomitant therapy with other investigational agents or participation in another clinical trial within 3 months of signature of ICF
10. Previous use of pentamidine with treatment discontinuation of less than 6 months prior to signature of ICF
11. Any of the following conditions: Ongoing clinically significant cardiac dysrhythmias such as atrial fibrillation ; QTc interval > 450 msec for males or > 470 msec for females or uncontrolled intercurrent cardiac illness, e.g. unstable angina; severe coronary disease, ventricular arrhythmias, bradycardia < 50 bpm (unless caused by beta-blocker); a history of additional risk factors for torsades de pointes (e.g., heart failure or family history of Long QTC Syndrome)
12. Presence of clinically significant hypokalemia or hypomagnesemia
13. Concurrent use of nephrotoxic drugs
14. Concurrent use of cardiotoxic drugs
15. Concurrent use of drugs that may be associated with pancreatitis
16. History of allergy or hypersensitivity to pentamidine
17. Pregnancy or breastfeeding. All female subjects of childbearing potential must have a negative urine pregnancy test prior to first dose of study medication.
18. Acute or chronic severe medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with trial participation of study drug administration, or which in the judgement of the investigator, would make the subject inappropriate for entry into this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 3 days
  Liver concentration of pentamidine in hepatocellular carcinoma tumor and surrounding tissue after oral administration for 3 days at different doses, measured in liver biopsies obtained during thermal ablation procedure

SECONDARY OUTCOMES:
plasma Pharmacokinetics | 3 days
  Plasma concentration of pentamidine after oral administration for 3 days at different doses
Adverse events | 3 days
  Safety as assessed by adverse events (AE), vital signs and laboratory parameters
markers of efficacy | 3 days
  The levels of Plasma pharmacodynamic markers of efficacy: ALT and AST
Biomarker | 3 days
  Tissue biomarker of mechanism of action: Endo-exonuclease

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Colin, B.Pharm, PhD, Study Director — Verlyx Pharma Inc
Locations (3):
- Canada (3):
  - Dr. Kelly Burak, Calgary, Alberta
  - Dr Morris Sherman, Toronto, Ontario
  - Dr Marc Bilodeau, Montreal, Quebec